CLINICAL TRIAL: NCT02246517
Title: The Effect of N2O on Chronic Neuropathic Pain
Brief Title: The Effect of N2O on Chronic Neuropathic Pain Patients
Acronym: N2O
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, michal roll, Dr, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TASMC-14-SB-0318-CTIL
Record Dates: First submitted 2014-07-15; First posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- N2O&Oxygen (Experimental): 70% N2O & 30% Oxygen by Aspiration for 5 min
  Interventions: Drug: N2O
- Oxygen (Placebo Comparator): 100% Oxygen by Aspiration for 5 min
  Interventions: Drug: Oxygen

INTERVENTIONS:
Drug: N2O
  Arms: N2O&Oxygen
Drug: Oxygen
  Arms: Oxygen

SUMMARY:
Important pharmacological agents for treatment of chronic neuropathic pain such as ketamine block NMDA receptors. Nitrous oxide, an inhalant agent used extensively In anesthesia, also have antagonist property of NMDA receptors. The investigators hypothesize that prolonged treatment with N2O can alleviate chronic neuropathic pain of different causes (e.g. diabetic neuropathy, post herpetic neuralgia etc.).

DETAILED DESCRIPTION:
Important pharmacological agents for treatment of chronic neuropathic pain such as ketamine block NMDA receptors. Nitrous oxide, an inhalant agent used extensively In anesthesia, also have antagonist property of NMDA receptors. The investigators hypothesize that prolonged treatment with N2O can alleviate chronic neuropathic pain of different causes (e.g. diabetic neuropathy, post herpetic neuralgia etc.). In order to examine our theory we Will recruit 40 patients aged 18-65 that suffer from chronic neuropathic pain. The patients will be divided to two groups of which half will receive treatment with N2O and half with placebo (pure O2) as a repeated weekly treatment for 4 weeks. At the beginning of the each session the patient will be asked to fill questionnaires regarding their pain quality and severity

ELIGIBILITY:
Inclusion Criteria:

* men and women at the age 18-65
* patient that suffer from chronic neuropathic pain
* VAS>40
* DN4 score >4
* takes pain medication on a regular basis
* Didn't get epidural injection for the pas month
* signed an informed consent form

Exclusion Criteria:

* patients that suffer from chronic lung disease.
* patients with cancer
* patients with heart disease
* pregnant and lactate woman
* patients that suffer from depression

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
change in adult pain as measured by visual Analog Scale for Pain (VAS Pain) | baseline and average of week for 4 weeks
  Assessment of pain in the last 24 hours before the visit by VAS

SECONDARY OUTCOMES:
change in adult pain as measured by Short-Form McGill Pain Questionnaire (SF-MPQ) | baseline and average of week for 4 weeks
  Assessment of pain in the last 24 hours before the visit by SF-MPQ

CONTACTS AND LOCATIONS:
Locations (1):
- Pain Medicine Unit, Tel Aviv, Israel